CLINICAL TRIAL: NCT04291638
Title: Evaluating an Online Adjunctive Support Following Intensive Services (OASIS) Strategy for Youth With Selective Mutism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-0010
Record Dates: First submitted 2020-02-21; First posted 2020-03-02 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Selective Mutism
MeSH Terms: conditions — Mutism

STUDY DESIGN:
Intervention Model Description: All participating families attend videoconferencing-based group parent training sessions. Families are given the opportunity to opt in to participate in the videoconferencing-based intensive group behavioral treatment program (remote IGBT).
Who Masked: Outcomes Assessor
Masking Description: "Independent evaluators" assigned to assess outcomes at Post-IGBT and School Year Follow-Up time points will be unfamiliar with families' progress during the IGBT, as well as masked to treatment participation (i.e., whether or not families participated in the remote IGBT).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Caregiver Training (Experimental): The Remote Caregiver Training arm consists of participation in a 5-hour, videoconferencing-based caregiver training program.
  Interventions: Behavioral: Remote Caregiver Training
- Remote Caregiver Training + Intensive Treatment (Experimental): The Remote Caregiver Training + Intensive Treatment arm consists of participation in a 5-hour, videoconferencing-based caregiving training program, followed by participation in the videoconferencing-based intensive group behavioral treatment program.
  Interventions: Behavioral: Remote Caregiver Training; Behavioral: Remote Intensive Group Behavioral Treatment (IGBT)

INTERVENTIONS:
Behavioral: Remote Caregiver Training — The remote caregiver training is a 5-hour videoconferencing-based training program that focuses on teaching cognitive behavioral therapy skills to the caregivers of children with selective mutism in a group format across 3 sessions.
Behavioral: Remote Intensive Group Behavioral Treatment (IGBT) — The remote IGBT is a 5-day videoconferencing-based treatment program that delivers cognitive behavioral therapy to children and their caregivers in a group format across 2-3 hours per day.
  Arms: Remote Caregiver Training + Intensive Treatment

SUMMARY:
This study sought to evaluate an innovative post-acute continuation/transition planning treatment strategy that leveraged an in-person intensive treatment followed by online, videoconferencing-based "booster" sessions for youth with selective mutism (SM). Twenty children between the ages of 4 and 10 and their caregivers were scheduled to participate in an in-person intensive group behavioral treatment (IGBT) for SM and subsequently randomized to receive either (a) six, biweekly, hour-long, videoconferencing-delivered booster sessions or (b) no additional treatment for 12 weeks. Due to COVID-19-related physical distancing restrictions, the study team was unable to provide in-person services. Thus, the clinical trial was converted to an open-trial design focused on evaluating remote treatment options (i.e., remotely delivered caregiver training sessions and/or a remotely delivered IGBT) for these families. All families retained in the study have or will participate(d) in assessments at the following time points: Intake (i.e., 4-5 months prior to the remote IGBT); Baseline (i.e., 1 month prior to the IGBT), Post-IGBT (i.e., 2 weeks following the IGBT), and School Year Follow Up (i.e., 16 weeks following the IGBT).

ELIGIBILITY:
Inclusion Criteria:

* Child between the ages of 4-10 years, and his or her caregiver(s)
* Child meets DSM-5 criteria for selective mutism diagnosis
* Child speaks English fluently

Exclusion Criteria:

* Child is identified as having any psychiatric condition significantly more impairing than selective mutism that requires alternate treatment
* The child is nonverbal with all caregivers

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions - Improvement (CGI-I) Scale rating at Post-IGBT | Up to 3 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The CGI-I Scale (Guy & Bonato, 1970) is a widely used global improvement measure; improvement is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Independent evaluators masked to family participation/progress during the intensive group behavioral treatment (IGBT) will complete the CGI-I rating. "Treatment Response" is defined as an independent evaluator rated CGI-I rating of 1 or 2 (ratings >/= 3 represent "Treatment Nonresponse").
Clinical Global Impressions - Improvement (CGI-I) Scale rating at School Year Follow Up | 16-18 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The CGI-I Scale (Guy & Bonato, 1970) is a widely used global improvement measure; improvement is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Independent evaluators masked to family participation/progress during the intensive group behavioral treatment (IGBT) and the post-acute strategy will complete the CGI-I rating. "Treatment Response" is defined as an independent evaluator rated CGI-I rating of 1 or 2 (ratings >/= 3 represent "Treatment Nonresponse").

SECONDARY OUTCOMES:
Change from Baseline in Anxiety Disorders Interview Schedule for Children (ADIS) Clinical Severity Ratings (CSRs) at Post-IGBT | Up to 3 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The ADIS (Silverman & Albano, 1996) is a well-supported semi-structured diagnostic interview assessing child mental disorders in accordance with the Diagnostic and Statistical Manual (DSM). Disorders are assigned a clinical severity rating (CSR) along a 9-point scale ranging from 0-8 (CSRs >/= 4 indicate diagnostic criteria were met). Independent evaluators masked to family participation/progress during the caregiver training program and/or intensive group behavioral treatment (IGBT) will administer the ADIS and determine CSRs.
Change from Baseline in Anxiety Disorders Interview Schedule for Children (ADIS) Clinical Severity Ratings (CSRs) at School Year Follow Up | 16-18 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The ADIS (Silverman & Albano, 1996) is a well-supported semi-structured diagnostic interview assessing child mental disorders in accordance with the Diagnostic and Statistical Manual (DSM). Disorders are assigned a clinical severity rating (CSR) along a 9-point scale ranging from 0-8 (CSRs >/= 4 indicate diagnostic criteria were met). Independent evaluators masked to family participation/progress during the caregiver training program and/or intensive group behavioral treatment (IGBT) and post-acute strategy will administer the ADIS and determine CSRs.
Change from Post-IGBT in Anxiety Disorders Interview Schedule for Children (ADIS) Clinical Severity Ratings (CSRs) at School Year Follow Up | 16-18 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The ADIS (Silverman & Albano, 1996) is a well-supported semi-structured diagnostic interview assessing child mental disorders in accordance with the Diagnostic and Statistical Manual (DSM). Disorders are assigned a clinical severity rating (CSR) along a 9-point scale ranging from 0-8 (CSRs >/= 4 indicate diagnostic criteria were met). Independent evaluators masked to family participation/progress during the caregiver training program and/or intensive group behavioral treatment (IGBT) will administer the ADIS and determine CSRs.
Change from Baseline in Children's Global Assessment Scale (CGAS) rating at Post-IGBT | Up to 3 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The CGAS (Shaffer et al., 1983) is a widely used measure of overall child disturbance, with scores ranging from 0-100. Lower scores indicate greater functional impairment. Independent evaluators masked to family participation/progress during the caregiver training program and/or intensive group behavioral treatment (IGBT) will complete the CGAS rating.
Change from Baseline in Children's Global Assessment Scale (CGAS) rating at School Year Follow Up | 16-18 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The CGAS (Shaffer et al., 1983) is a widely used measure of overall child disturbance, with scores ranging from 0-100. Lower scores indicate greater functional impairment. Independent evaluators masked to family participation/progress during the caregiver training program and/or intensive group behavioral treatment (IGBT) will complete the CGAS rating.
Change from Post-IGBT in Children's Global Assessment Scale (CGAS) rating at School Year Follow Up | 16-18 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The CGAS (Shaffer et al., 1983) is a widely used measure of overall child disturbance, with scores ranging from 0-100. Lower scores indicate greater functional impairment. Independent evaluators masked to family participation/progress during the caregiver training program and/or intensive group behavioral treatment (IGBT) will complete the CGAS rating.
Change from Baseline in Selective Mutism Questionnaire (SMQ) scores at Post-IGBT | Up to 3 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The SMQ (Bergman et al., 2008) is a well-supported parent-report questionnaire with 23 items assessing child verbal behavior across settings (i.e., home, school, community) and associated impairment. Items are rated from 0 (never) to 3 (always).
Change from Baseline in Selective Mutism Questionnaire (SMQ) scores at School Year Follow Up | 16-18 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The SMQ (Bergman et al., 2008) is a well-supported parent-report questionnaire with 23 items assessing child verbal behavior across settings (i.e., home, school, community) and associated impairment. Items are rated from 0 (never) to 3 (always).
Change from Post-IGBT in Selective Mutism Questionnaire (SMQ) scores at School Year Follow Up | 16-18 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The SMQ (Bergman et al., 2008) is a well-supported parent-report questionnaire with 23 items assessing child verbal behavior across settings (i.e., home, school, community) and associated impairment. Items are rated from 0 (never) to 3 (always).
Change from Baseline in School Speech Questionnaire (SSQ) scores at School Year Follow Up | 16-18 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The SSQ (Bergman et al., 2002) is a teacher-report adapted from the SMQ with 6 items assessing child verbal behavior in school. Items are rated from 0 (never) to 3 (always).
Change from Baseline in Impairment Rating Scale - Parent Version (IRS-P) at School Year Follow Up | 16-18 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The IRS-P (Fabiano et al., 2006) is a 7-item parent-report measure of child impairment in the home, community, and school settings. Items are rated on a 7-point scale ranging from 0 (no problem) to 6 (extreme problem).
Change from Baseline in Impairment Rating Scale - Teacher Version (IRS-T) at School Year Follow Up | 16-18 weeks after the Intensive Group Behavioral Treatment (IGBT)
  The IRS-T (Fabiano et al., 2006) is an 8-item teacher-report measure of child impairment in the school setting. Items are rated on a 7-point scale ranging from 0 (no problem) to 6 (extreme problem).

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Hong, M.S., Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT04291638/ICF_001.pdf